CLINICAL TRIAL: NCT02593747
Title: A Single-dose, Single-center, Randomized, Open-label, Two-way Crossover Study in Healthy Adults to Assess the Bioequivalence of Loratadine Oral Solution/Syrup 1mg/mL (GPLA Formula) Versus Claritin Peach Syrup 1mg/mL (ANNA Formula)
Brief Title: To Assess Bioequivalence of Loratadine Oral Solution/Syrup Versus Claritin Peach Syrup
Acronym: Bordeaux
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 18199; 2015-002720-12 (EudraCT Number)
Record Dates: First submitted 2015-10-30; First posted 2015-11-02 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Histamine H1 Antagonists, Non-Sedating
Keywords: Allergy
MeSH Terms: conditions — Hypersensitivity | interventions — Loratadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Loratadine oral solution/syrup then Claritin peach syrup (Experimental): Subjects received a single oral dose of 10 mg loratadine-oral solution/syrup 1 mg/mL (GPLA formula, test formulation) under fasted condition in treatment period 1, followed by a single oral dose of 10 mg loratadine-claritin peach syrup 1 mg/mL (ANNA formula, reference formulation) under fasted condition in treatment period 2. A wash-out period of at least 10 calendar days was maintained between the 2 treatments.
  Interventions: Drug: Loratadine oral solution; Drug: Loratadine (Claritin peach syrup)
- Claritin peach syrup then Loratadine oral solution/syrup (Experimental): Subjects received a single oral dose of 10 mg loratadine-claritin peach syrup 1 mg/mL (ANNA formula, reference formulation) under fasted condition in treatment period 1, followed by a single oral dose of 10 mg loratadine-oral solution/syrup 1 mg/mL (GPLA formula, test formulation) under fasted condition in treatment period 2. A wash-out period of at least 10 calendar days was maintained between the 2 treatments.
  Interventions: Drug: Loratadine oral solution; Drug: Loratadine (Claritin peach syrup)

INTERVENTIONS:
Drug: Loratadine oral solution — Subjects received a single oral dose of 10 mg loratadine oral solution/syrup 1 mg/mL (GPLA formula, test formulation) under fasted condition in any intervention period.
Drug: Loratadine (Claritin peach syrup) — Subjects received a single oral dose of 10 mg loratadine claritin peach syrup 1 mg/mL (ANNA formula, reference formulation) under fasted condition in any intervention period.

SUMMARY:
To assess the bioequivalence of Loratadine Oral Solution/Syrup 1mg/mL (GPLA Formula) versus Claritin Peach Syrup 1mg/mL (ANNA Formula)

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult (men or women), age 18 to 55 years inclusive;
* Body mass index 18.5 to 30.0 kg/m*2 inclusive;
* Able to read and understand the written informed consent for study-related information and instruction;
* Able to comply with protocol requirements, including overnight stays, blood sample collections as defined in the protocol;
* Agree not to donate whole blood or components of blood (e.g. plasma, thrombocytes) starting from signing the informed consent form through 30 days after the last study procedure, except for the blood samples collected for this study;
* Female subjects of childbearing potential must be using a medically acceptable form of birth control for at least 1 month prior to screening (3 months on oral contraceptives), e.g., oral or patch contraceptives, intrauterine device, injectable contraceptive (e.g. Depo-Provera), or a double barrier and have a negative pregnancy test at Screening and prior to study drug administration on Day 0 of Dosing Periods 1 and 2. Female subjects of non-childbearing potential must be amenorrheic for at least two years or had a hysterectomy and/or bilateral oophorectomy;

Exclusion Criteria:

* Pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study drugs will not be normal;
* Known hypersensitivity to any medication (active substances or excipients of the preparations) to be used in the study;
* Known galactose intolerance, lactase deficiency or glucose-galactose malabsorption
* Known severe allergies (e.g. allergies to more than 3 allergens, allergies affecting the lower respiratory tract - allergic asthma, allergies requiring therapy with corticosteroids);
* Use of, within 1 month before the first study drug administration, systemic or topical medicines or substances which might affect the study objectives, e.g

  * any drug known to induce cytochrome P3A4/5 or P Glycoprotein (e.g. rifampin, carbamazepine, St. John's wort);
  * any drug known to inhibit cytochrome P3A4/5 or P Glycoprotein (e.g. erythromycin, clarithromycin, chloramphenicol, ketoconazole);
  * any drug known to induce cytochrome P2D6 (e.g. rifampin, dexamethasone);
  * any drug known to inhibit cytochrome P2D6 (e.g. cimetidine, desipramine, fluoxetine, metoclopramide);
* Positive urine pregnancy, urine drug test or Hepatitis B, hepatitis C or HIV tests;
* Clinically relevant findings in the physical examination, e.g., signs of bleeding diathesis, signs of heart failure, evidence of peripheral circulatory disturbances, and skin abnormalities;

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2015-12; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Primary: Area Under the Concentration Versus Time Curve From Zero to the Last Data Point Greater Than Lower Limit of Quantitation (LLOQ) of Loratadine in Plasma (AUC[0-tlast]) After Single Oral Dose of Loratadine | 0 hour (h) (pre-dose) to 72 h post-dose
  Area under the concentration versus time curve from zero to the last data point greater than (>) LLOQ (AUC[0-tlast]) after single dose.
Maximum Observed Concentration (Cmax) of Loratadine in Plasma After Single Oral Dose of Loratadine | 0 h (pre-dose) to 72 h post-dose
  Maximum observed loratadine concentration in plasma, directly taken from analytical data.

SECONDARY OUTCOMES:
Time to Reach Maximum Concentration (tmax) in Plasma After Single Dose of Loratadine | 0 h (pre-dose) to 72 h post-dose
  Time to reach maximum loratadine concentration in plasma after its single oral dose, directly taken from analytical data.
Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC) of Loratadine in Plasma After Single Dose | 0 h (pre-dose) to 72 h post-dose
  Area under the concentration versus time curve from zero to infinity after single dose.
Half-Life (t1/2) Associated With the Terminal Slope of Loratadine After Single Dose | 0 h (pre-dose) to 72 h post-dose
  Half-life associated with the terminal slope.
Total Body Clearance (CL/F) of Loratadine Calculated After its Single Oral Administration | 0 h (pre-dose) to 72 h post-dose
  Total body clearance of loratadine calculated after extravascular application.
Percentage of Area Under the Concentration Versus Time Curve (AUC) From the Last Calculated Data Point Greater Than Lower Limit of Quantification [LLOQ]) to Infinity (%AUC[tlast-∞]) After Single Oral Administration of Loratadine | 0 h (pre-dose) to 72 h post-dose
  Percentage of AUC from the last calculated data point > LLOQ to infinity was measured.
Apparent Terminal Rate Constant (λz) of Loratadine After Single Dose | 0 h (pre-dose) to 72 h post-dose
  Apparent terminal rate constant, calculated from the slope of a log-linear regression of the unweighted data considering the last concentration-time points > LLOQ.
Area Under the Concentration Versus Time Curve From Zero to 72 Hours (AUC[0-72]) of Lloratadine in Plasma After Single Oral Dose | 0 h (pre-dose) to 72 h post-dose
  Area under the concentration versus time curve from zero to 72 h after single dose.
Maximum Observed Concentration (Cmax) of Desloratadine in Plasma After Single Oral Dose of Loratadine | 0 h (pre-dose) to 72 h post-dose
  Maximum observed desloratadine concentration in plasma, directly taken from analytical data.
Time to Reach Maximum Concentration (tmax) of Desloratadine in Plasma After Single Dose of Loratadine | 0 h (pre-dose) to 72 h post-dose
  Time to reach maximum drug concentration in the measured matrix, directly observed from the analytical data.
Area Under the Concentration Versus Time Curve From Zero to the Last Data Point Greater Than Lower Limit of Quantitation (LLOQ) of Desoratadine in Plasma (AUC[0-tlast]) After Single Oral Dose of Loratadine | 0 h (pre-dose) to 72 h post-dose
  Area under the concentration versus time curve from zero to the last data point > LLOQ (AUC[0-tlast]) after single dose.
Area Under the Concentration Versus Time Curve From Zero to 72 Hours (AUC[0-72]) of Desloratadine in Plasma After Single Oral Dose of Loratadine | 0 h (pre-dose) to 72 h post-dose
  Area under the concentration versus time curve from zero to 72 h after single dose. AUC and residual area were not evaluated because the concentration at 72 h was quantifiable in the majority of profiles.
Time of Last Concentration Above the Lower Limit Of Quantitation (LLOQ) of Desloratadine, Directly Taken From Analytical Data (tlast) | 0 h (pre-dose) to 72 h post-dose
  Time of last concentration above LLOQ, directly taken from analytical data.
Half-Life (t1/2) Associated With the Terminal Slope of Desoratadine After Single Dose of Loratadine | 0 h (pre-dose) to 72 h post-dose
  Half-life associated with the terminal slope.
Percentage of Area Under the Concentration Versus Time Curve (AUC) from the Last Data Point Greater Than Lower Limit of Quantitation (LLOQ) to Infinity (%AUC[tlast-∞]) of Desoratadine After Single Oral Administration of Loratadine | 0 h (pre-dose) to 72 h post-dose
  Percentage of area under the concentration versus time curve from zero to the last data point > LLOQ in plasma (AUC[(0-tlast]) was measured.
Apparent Terminal Rate Constant (λz) of Desoratadine After Single Dose of Loratadine | 0 h (pre-dose) to 72 h post-dose
  Apparent terminal rate constant, calculated from the slope of a log-linear regression of the unweighted data considering the last concentration-time points > LLOQ.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Neu-Ulm, Bavaria, Germany

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/